CLINICAL TRIAL: NCT01542697
Title: Phase IV Recruiting
Brief Title: Effect of Intraperitoneal Nebulisation of Magnesium Sulphate for Analgesia Following Laparoscopic Cholecystectomy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: B.P. Koirala Institute of Health Sciences (Other)
Responsible Party: Principal Investigator, sujata niroula, junior resident, B.P. Koirala Institute of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 698/067/068
Record Dates: First submitted 2012-02-27; First posted 2012-03-02 (Estimated); Last update posted 2012-03-02 (Estimated); Status verified 2012-02

CONDITIONS: Postoperative Pain
Keywords: magnesium sulpahate; postoperative analgesia
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Magnesium sulphate (Active Comparator): intraperitoneal nebulisation of 1.5 gm of magnesium sulphate with 2 ml of normal saline at the end of surgery before closure
  Interventions: Drug: intraperitoneal nebulisation of magnesium sulphate
- normal saline (Placebo Comparator): intraperitoneal nebulisation of 5 ml of normal saline after end of surgery before closure
  Interventions: Drug: intraperitoneal nebulisation of magnesium sulphate

INTERVENTIONS:
Drug: intraperitoneal nebulisation of magnesium sulphate — intraperitoneal nebulisation of 1.5 gm of magnesium sulphate with 2 ml of normal saline

SUMMARY:
intraperitoneal nebulisation with magnesuim sulphate will reduce post operative pain and analgesic consumption in postoperative period following laparoscopic cholecystectomy.

DETAILED DESCRIPTION:
Sixty patients undergoing laparoscopic cholecystectomy belonging to American Society of Anaesthesiologist (I-II) of age 18-65 yrs will be enrolled.Group one (n=30) will receive 1.5 gm magnesium sulphate diluted in 3ml of normal saline and group 2 (n=30) will receive 5 ml of NS.

ELIGIBILITY:
Inclusion Criteria: ASA I-II

-

Exclusion Criteria: history of

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
number of analgesic request | 24 hour
  time to first analgesic request is taken as duration of effective analgesia
  number of analgesic request in first 24 hours were also counted

SECONDARY OUTCOMES:
VAS score | first complaint of pain, 6 hrs, 12 hrs, 24 hrs
  Visual analogue scale is a linear 10cm scale with 0 corresponding to no pain and 10 to worst pain ever
nausea and vomiting | 24 hrs
respiratory rate | 24 hrs
sedation | 24hrs

CONTACTS AND LOCATIONS:
Overall Officials: krishna Pokharel, MD, Study Director — B.P. Koirala Institute of Health Sciences
Locations (1):
- routine operation theatre of BPKoirala, Dharān, Nepal

REFERENCES:
- [Background] Alkhamesi NA, Peck DH, Lomax D, Darzi AW. Intraperitoneal aerosolization of bupivacaine reduces postoperative pain in laparoscopic surgery: a randomized prospective controlled double-blinded clinical trial. Surg Endosc. 2007 Apr;21(4):602-6. doi: 10.1007/s00464-006-9087-6. Epub 2006 Dec 16. PMID 17180268
- [Background] Abdel - Raouf M, Amer H. Postoperative analgesic effects of intraperitoneal NMDA receptor antagonist (ketamine and magnesium sulphate )in patients undergoing laparoscopic cholecystectomy .Eg J Anaesth. 2004;20: 107-11